CLINICAL TRIAL: NCT00728169
Title: Feasibility of Developing an Effective Asthma Intervention Using CBPR Methods
Brief Title: Developing Asthma Interventions Using Community Based Research
Status: Completed | Type: Observational
Sponsor: Meharry Medical College (Other)
Responsible Party: David Scott Trochtenberg, M.D., Meharry Medical College
Other Study IDs: 020715JEM13314; P20RR011792 (NIH)
Record Dates: First submitted 2008-07-31; First posted 2008-08-05 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Asthma
Keywords: Asthma; Focus Group; Community Based Participatory Research
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to identify community resources and challenges in improving the health of community members with asthma.

The primary goal of this project is to use Community-Based Participatory Research methodology to develop interventions aimed at improving asthma management in high-risk African American asthmatics. This "ground-up" longterm approach has never been tested before in asthmatics. The primary goal of this study will be accomplished with four specific aims:

Aim 1. Conduct focus groups to identify barriers to asthma management in the target population.

Aim 2. Use a community advisory board (CAB) consisting of participants selected from the various focus groups to gather information about solutions for the above barriers.

Aim 3. Use the information from the CAB to develop an intervention to improve asthma self management behaviors in the target population.

Aim 4. Refine the developed intervention based on feedback from focus groups conducted in Aim 1.

DETAILED DESCRIPTION:
Volunteer will be asked to respond to several questions that address their perceptions about asthma. Volunteers will also be asked to discuss their beliefs about asthma. Everyone in the group will be given an opportunity to answer questions. Volunteers can decide that they no longer want to participate in the group discussion at any time.

The discussion will last from 1.5 - 2 hours. The focus group discussion will have a maximum of 10 people.

We will be audio and video taping the discussion so that we do not miss any information that volunteers share with us. The audio and video tapes will not be shared with anyone outside our staff.

Volunteer participation in this study is voluntary and there will be no negative consequences if volunteers decide not to participate. Volunteers are also free to withdraw from this study at any time. Withdrawal or refusal to participate will not affect health care services or other rights.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African-American, 18 yrs. or older, resident of Davidson County, Tennessee at least 1 year.

Exclusion Criteria:

* Under 18 yrs. of age
* Non-African American
* Non-English speaking
* Do not reside in Davidson County, Tennessee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African-American, 18 years and older
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2008-07; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Use information from Community Based Participatory Research to develop an intervention to improve asthma self management behaviors. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David S Trochtenberg, MD, Principal Investigator — Meharry Medical College
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States